CLINICAL TRIAL: NCT00620204
Title: Efficacy Study of Atorvastatin to Treat Variant Angina
Acronym: ESAVA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: HC Gwon, MD,PhD / Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-01-018
Record Dates: First submitted 2008-02-10; First posted 2008-02-21 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Angina Pectoris, Variant
Keywords: atorvastatin; Angina Pectoris, Variant; endothelial dysfunction
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Atorvastatin group
  Interventions: Drug: atorvastatin
- B (No Intervention): Control group

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 40mg qd for 1 year
  Other Names: Lipitor®
  Arms: A

SUMMARY:
The objective of this study is to evaluate effect of statin treatment for vasospastic angina.

DETAILED DESCRIPTION:
Vasospastic angina is presented by myocardial ischemia with spasm of coronary artery accompanying chest pain or discomfort. The precise mechanisms have not been established, but a reduction in NO (nitric oxide) production, an imbalance between endothelium-derived relaxing and contracting factors,or an injury of endothelium have been suggested.

Impaired FMD(flow mediated endothelium-dependent vasodilation) in the brachial artery was demonstrated in vasospastic angina,and improvement of endothelial dysfunction with treatment of statin is documented in several studies.

So, we expect that statin treatment for vasospastic angina provide additional therapeutic effects via improvement of endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Vasospastic angina or spontaneous spasm during coronary angiography (Vasospastic angina is defined as Thrombolysis In Myocardial Infarction (TIMI) flow grade 0-2 noted in intracoronary ergonovine provocation test and development of chest pain or EKG change; Spontaneous spasm is defined as TIMI flow grade 0-2 of coronary artery without ergonovine injection)
* Normal or insignificant lesion (diameter stenosis <50%) on coronary angiography

Exclusion Criteria:

* Elevated liver enzyme: serum aspartate aminotransferase or alanine aminotransferase concentrations more than 3 times the upper limit of normal
* Significant lesion( diameter stenosis ≥50%) documented in coronary angiography
* Pregnancy
* Prior percutaneous coronary intervention or coronary artery bypass surgery
* Previous statin use
* Impaired renal function with serum creatinine ≥ 2.0 mg/dl
* Severe left ventricular dysfunction ( LVEF ≤ 30% on echocardiography)
* Myopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Ergonovine provocation test 24hrs later after admission | 1 year later

SECONDARY OUTCOMES:
Chest pain with EKG change during admission for 24hrs at 12mo. later (All medications are withheld for 48hrs. before admission) | 1year later

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-chul Gwon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea